CLINICAL TRIAL: NCT05030857
Title: An Open-label, Fixed Sequence, Drug-drug Interaction Study in Healthy Subjects to Evaluate the Effect of GLPG4716 on the Pharmacokinetics of Midazolam, a Sensitive Index Substrate of CYP3A4, and to Assess the Effect of Food on the Pharmacokinetics of GLPG4716
Brief Title: Drug-drug Interaction and Food-effect Study With GLPG4716 and Midazolam in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GLPG4716-CL-102
Record Dates: First submitted 2021-08-30; First posted 2021-09-01 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GLPG4716 and Midazolam (Experimental)
  Interventions: Drug: GLPG4716; Drug: Midazolam

INTERVENTIONS:
Drug: GLPG4716 — From Day 3 to Day 14, participants will receive GLPG4716 tablets once daily in fasted state. On Day 8 GLPG4716 will be administered in fed state.
Drug: Midazolam — On Days 1, 3 and 13, participants will receive a single oral dose of MDZ as an oral solution in fasted state.

SUMMARY:
The purpose of this study is to determine the effect of the administration of multiple doses of GLPG4716 on the amount of midazolam (MDZ) that gets into the blood when the two drugs are administered together compared to when midazolam is administered alone. Other objectives of this study are to evaluate the safety and tolerability of GLPG4716 when administered with midazolam and assess the amount of GLPG4716 that gets into the blood when administered with midazolam. This study will also assess the effect of food on the amount of GLPG4716 that gets into the blood.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 55 years of age (extremes included), on the date of signing the informed consent form. Female subjects should be of non-childbearing potential.
* A body mass index between 18.0 and 30.0 kg/m2, inclusive.
* Judged to be in good health by the investigator based upon:

  * The results of a medical history
  * Physical examination
  * Vital signs
  * Oxygen saturation
  * 12-lead electrocardiogram
  * Fasting clinical laboratory safety tests. Aspartate aminotransferase and alanine aminotransferase must be no greater than 1.5x upper limit of normal range and total bilirubin no greater than 1x upper limit of normal. Other clinical laboratory safety test results must be within the reference ranges or test results that are outside the reference ranges need to be considered not clinically significant in the opinion of the investigator.

This list only contains the key inclusion criteria.

Exclusion Criteria:

* Known hypersensitivity to ingredients of GLPG4716 and/or MDZ
* History of a significant allergic reaction to ingredients of GLPG4716 and/or MDZ as determined by the investigator.
* Treatment with any medication including:

  * Over-the-counter and/or prescription medication
  * Dietary supplements
  * Nutraceuticals, vitamins and/or herbal supplements, and hormonal replacement therapy
  * Except occasional paracetamol (maximum dose of 2 g/day and maximum of 10 g/2 weeks) in the last 2 weeks or 5 half-lives of the drug, whichever is longer, prior to the first dosing.

This list only contains the key exclusion criteria.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2021-11-13 (Actual); Study Completion 2021-11-13 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of MDZ | From Day 1 pre-dose until Day 15
  To determine the effect of GLPG4716 on the pharmacokinetics (PK) of MDZ
Area under the plasma concentration-time curve from time zero to infinity (AUC0-inf) of MDZ | From Day 1 pre-dose until Day 15
  To determine the effect of GLPG4716 on the PK of MDZ

SECONDARY OUTCOMES:
Cmax of GLPG4716 | From Day 1 pre-dose until Day 15
  To assess the effect of food on the PK of GLPG4716.
Area under the plasma concentration-time curve over the dosing interval (AUCt) of GLPG4716 | From Day 1 pre-dose until Day 15
  To assess the effect of food on the PK of GLPG4716.
Frequency and severity of treatment-emergent adverse events (TEAEs), treatment-emergent (SAEs), and TEAEs leading to treatment discontinuations | From Day 1 through study completion, an average of one month
  To evaluate the safety and tolerability of GLPG4716 when co-administered with MDZ

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Rueda-Rincon, MD, Study Director — Galapagos NV
Locations (1):
- Altasciences, Montreal, Canada

IPD SHARING:
Plan to Share IPD: No